CLINICAL TRIAL: NCT02541825
Title: Using Covered Stent of Diameter of 7mm in a Prospective, Single Blind, Randomized, Controlled Study of TIPS(Transjugular Intrahepatic Portosystemic Stent Shunt )
Brief Title: Using Covered Stent of Diameter of 7mm in TIPS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Shijitan Hospital, Capital Medical University (Other)
Responsible Party: Principal Investigator, Fuquan Liu, Director,Clinical Research, Beijing Shijitan Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BeijingShijitan
Record Dates: First submitted 2015-09-03; First posted 2015-09-04 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Liver Disease
Keywords: transjugular intrahepatic portosystemic shunt
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the stent of diameter of 7mm (Experimental): Procedure/Surgery:Jugular vein puncture and catheterization. Device:RUPS-100(COOK Company)sheath ,7mm balloon,Pigtail catheter,the stent of diameter of 7mm (Bard,Fluency) Drug(including placebo):No Biological/Vaccine:No
  Interventions: Device: the stent of diameter of 7mm
- the stent of diameter of 8mm (Other): Procedure/Surgery:Jugular vein puncture and catheterization. Device:RUPS-100(COOK Company)sheath ,8mm balloon,Pigtail catheter,the stent of diameter of 8mm (Bard,Fluency) Drug(including placebo):No Biological/Vaccine:No
  Interventions: Device: the stent of diameter of 8mm

INTERVENTIONS:
Device: the stent of diameter of 7mm — 108 patients use the stent of diameter of 7mm in TIPS
  Arms: the stent of diameter of 7mm
Device: the stent of diameter of 8mm — 108 patients use the stent of diameter of 8mm in TIPS
  Arms: the stent of diameter of 8mm

SUMMARY:
This study evaluates the incidence of hepatic encephalopathy between covered stent of diameter of 7mm and 8mm in TIPS(transjugular intrahepatic portosystemic stent shunt ).Half of the participants will receive stent of diameter of 7mm ,while the other half will receive stent of diameter of 8mm.

DETAILED DESCRIPTION:
TIPS is effective in the treatment of hemorrhage of digestive tract and intractable ascites,which are the complications of cirrhosis. At present, the high incidence of hepatic encephalopathy has been a major problem after TIPS. The high incidence rate of hepatic encephalopathy was closly associated with the diameter of the stent. We often use the stent of diameter 8mm in TIPS.In this study, we try to use the stent of smaller diameter of 7mm in TIPS,and compare the incidence of hepatic encephalopathy between the stent of diameter of 7mm and 8mm .

ELIGIBILITY:
Inclusion Criteria:

1. there is a clear TIPS treatment indications of liver cirrhosis portal hypertension patients of gastrointestinal bleeding.
2. undergoing elective TIPS to treat patients.
3. aged 18-70 years old

Exclusion Criteria:

1. preoperative patients with hepatic encephalopathy.
2. with portal vein thrombosis patients.
3. combined liver malignant tumor or other parts of the patients with malignant tumor.
4. In combination of peptic ulcer bleeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of hepatic encephalopathy after TIPS | 1 year
  The incidence of hepatic encephalopathy after TIPS in 7day,1,3,6,12month

SECONDARY OUTCOMES:
the incidence of shunt restenosis after TIPS | 1 year
  The incidence of shunt restenosis after TIPS in 7day,1,3,6,12month
the recurrence rate of gastrointestinal bleeding after TIPS | 1 year
  The recurrence rate of gastrointestinal bleeding after TIPS in 7day,1,3,6,12month
Portal venous pressure before and afterTIPS | 1 year
  Portal venous pressure before and afterTIPS.
liver function in different periods | 1 year
  liver function during different periods before and after TIPS in 7day,1,3,6,12month
blood ammonia in different periods | 1 year
  blood ammonia before and after TIPS in 7day,1,3,6,12month
jaundice index in different periods | 1 year
  jaundice index before and after TIPS in 7day,1,3,6,12month
platelet count in different periods | 1 year
  platelet count before and after TIPS in 7day,1,3,6,12month

CONTACTS AND LOCATIONS:
Overall Officials: Jianli Xu, MD PhD, Study Chair — Beijing Shijitan Hospital, Capital Medical University